CLINICAL TRIAL: NCT00024336
Title: Treatment of Children With Newly Diagnosed Diffuse Pontine Gliomas Using Conventional Radiotherapy and High Dose Tamoxifen
Brief Title: Radiation Therapy and Tamoxifen in Treating Children With Newly Diagnosed Brain Stem Glioma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Children's Cancer and Leukaemia Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CCLG-CNS-1999-06; CDR0000068920 (Registry Identifier: PDQ (Physician Data Query)); EU-20123
Record Dates: First submitted 2001-09-13; First posted 2003-01-27 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2006-12

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: untreated childhood brain stem glioma
MeSH Terms: conditions — Central Nervous System Neoplasms | interventions — Tamoxifen; Radiotherapy

INTERVENTIONS:
Drug: tamoxifen citrate
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Tamoxifen may kill tumor cells by blocking the enzymes necessary for cell growth. Combining radiation therapy with tamoxifen may be effective in treating newly diagnosed brain stem glioma.

PURPOSE: Phase II trial to study the effectiveness of combining radiation therapy and tamoxifen in treating children who have newly diagnosed brain stem glioma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether high-dose tamoxifen with radiotherapy increases the median survival and overall survival of children with newly diagnosed brain stem gliomas.
* Determine the time to neurologic or radiographic progression in patients treated with this regimen.
* Determine the acute and chronic toxicity of high-dose tamoxifen in these patients.

OUTLINE: This is a multicenter study.

Patients undergo radiotherapy once daily 5 days a week for 6 weeks. Within 2 weeks after the initiation of radiotherapy, patients receive oral high-dose tamoxifen once daily. Tamoxifen continues in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: Approximately 60 patients will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Newly diagnosed tumor of the brain stem (diffuse intrinsic lesion centered on the pons)

  * Radiological and clinical diagnostic criteria allowed (biopsy not required)
  * The following astrocytic tumors are allowed if histologically confirmed:

    * Diffuse astrocytoma (all subtypes)
    * Anaplastic astrocytoma
    * Glioblastoma
    * Pilocytic astrocytoma (grade I)
* Less than 6 months since diagnosis
* At least 1 of the following signs of brain stem tumor:

  * Cranial nerve deficit
  * Long tract signs
  * Ataxia
* No focal lesions of the brain stem (either clearly marginated or cystic), cervicomedullary tumors, tumors predominately exophytic, or pontine tumors diagnosed as pilocytic on biopsy

PATIENT CHARACTERISTICS:

Age:

* Under 20

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* Not pregnant or nursing
* No frequent vomiting or other medical condition that would preclude oral medication intake

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy for brain stem glioma

Endocrine therapy:

* Concurrent steroids allowed

Radiotherapy:

* No prior radiotherapy for brain stem glioma

Surgery:

* Not specified

Other:

* Concurrent anticonvulsants allowed

Max Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 1999-08

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Michalski, MD, Study Chair — Great Ormond Street Hospital for Children NHS Foundation Trust
Locations (22):
- Our Lady's Hospital for Sick Children, Crumlin, Ireland
- United Kingdom (21):
  - Birmingham Children's Hospital, Birmingham, England
  - Bristol Royal Hospital for Children, Bristol, England
  - Addenbrooke's NHS Trust, Cambridge, England
  - St. James's Hospital, Leeds, England
  - Leicester Royal Infirmary, Leicester, England
  - Royal Liverpool Children's Hospital, Alder Hey, Liverpool, England
  - Saint Bartholomew's Hospital, London, England
  - Hospital for Sick Children NHS Trust, London, England
  - Middlesex Hospital- Meyerstein Institute, London, England
  - Manchester Children's Hospitals (NHS Trust), Manchester, England
  - Newcastle Upon Tyne Hospitals NHS Trust, Newcastle upon Tyne, England
  - Queen's Medical Centre, Nottingham, England
  - Oxford Radcliffe Hospital, Oxford, England
  - Children's Hospital - Sheffield, Sheffield, England
  - Southampton General Hospital, Southampton, England
  - Royal Marsden Hospital, Sutton, England
  - Royal Belfast Hospital for Sick Children, Belfast, Northern Ireland
  - Aberdeen Royal Infirmary, Aberdeen, Scotland
  - Royal Hospital for Sick Children, Edinburgh, Scotland
  - Royal Hospital for Sick Children, Glasgow, Scotland
  - Llandough Hospital, Penarth, Wales